CLINICAL TRIAL: NCT07145970
Title: Standardization of Spatial Neglect Assessment Tests in a Francophone Population
Brief Title: Standardization of Spatial Neglect Assessment Tests
Acronym: NOTEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP250520
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-07

CONDITIONS: Perceptual Disorders; Healthy Volunteers; Reference Values
Keywords: Spatial neglect; Tactile neglect; Visual neglect; Directional motor neglect
MeSH Terms: conditions — Perceptual Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group (Experimental)
  Interventions: Other: Neuropsychological assessment tests for spatial neglect

INTERVENTIONS:
Other: Neuropsychological assessment tests for spatial neglect — Standardized administration of four paper-and-pencil tests designed to assess different forms of spatial neglect:
  * Apples Cancellation Test (Birmingham Cognitive Screen) for egocentric and allocentric neglect,
  * Simplified Comb and Razor Test for personal and motor neglect,
  * Line Bisection Test (30 cm ruler, blind version) for tactile neglect,
  * Dot Test for visual exploration.
  The purpose is to establish normative reference scores in healthy French-speaking adults according to age, sex, and professional qualification. No therapeutic intervention or patient population is involved.

SUMMARY:
Spatial neglect is a common cognitive disorder in stroke patients, characterized by a lateralized deficit in attention and intention.

This research focuses on defining norms for tests to assess spatial neglect. The norms correspond to the results obtained in a population free of any disorder that could have an impact on test performance. These results can vary in a normal, non-pathological way, with certain parameters such as age, sex, laterality or level of education. Defining these norms in healthy volunteers is therefore essential for interpreting results in patients suspected of spatial neglect, and in particular for defining pathological thresholds above which the diagnosis of spatial neglect can be retained.

To answer the research question, we plan to include 210 people with no central neurological disease (stroke, epilepsy and multiple sclerosis in particular), in a single-center study in the neurovascular department of the Raymond-Poincaré hospital (Garches). The 210 subjects will be divided into 10-year age groups, from 20 to 89 years, with the recruitment of 30 participants per age group (15 men and 15 women): 20-29 years, 30-39 years, 40-49 years, 50-59 years, 60-69 years, 70-79 years, 80-89 years.

DETAILED DESCRIPTION:
Spatial neglect is a loss of attention to stimuli in the absence of sensory damage. It is most often a left egocentric hemineglect, due to involvement of the right perisylvian cortex, in which the patient neglects stimuli to his left. More recently, allocentric neglect has been described, where the patient neglects the right or left part of each stimulus. Egocentric neglect is common in stroke patients and correlates with poorer functional recovery and degraded quality of life. The prevalence and impact of allocentric neglect on patients is less well known, not least because of a lack of assessment tools. Tests have recently been developed in English to screen simultaneously for allocentric and egocentric visual neglect. These tests are based on target cancellation, such as whole or open apples in the Apples cancellation test of the Birmingham Cognitive Screen. There is currently no validated French-language version of these tests.

In the case of personal, motor and tactile neglect, these three components are difficult to separate. A patient's ability to indicate blindly, by tactile exploration, the middle of a ruler, or to explore by touch different targets placed in front of him/her, should, after standardization, enable exploration of these last two types of neglect. A simplified version of the Comb and Razor Test should enable assessment of personal and motor neglect.

The aim of this study is to establish mean scores for healthy French-speaking volunteers without central neurological disease on different spatial neglect assessment tests according to their age, sex and level of professional qualification, using French-translated instructions for taking and scoring the tests.

Healthy volunteers with no known history of stroke or cognitive impairment will be included prospectively in the neurovascular department of the Raymond-Poincaré hospital in Garches. We aim to recruit 30 subjects (15 men and 15 women) in 10-year age groups (20 to 29, 30 to 39, 40 to 49, 50 to 59, 60 to 69, 70 to 79 and 80 to 89), i.e. 210 subjects.

The significance threshold will be defined at 0.05. Statistical analyses will be performed using Rstudio software.

Qualitative variables will be described by their numbers and percentages, and quantitative variables by their means, standard deviations, minimums, maximums, as well as their medians and interquartile ranges (25th percentile - 75th percentile).

To identify the association between the variables (age, gender, level of qualification and laterality) and the metrics relating to the results of the following tests (Apples cancellation test, Comb and razor test, Peg test and Ruler blind bisection test) and their completion times, a linear regression will be conducted. The variables to be explained will be the metrics relating to the results of the following tests (Apple test, Comb and razor test, Plot test and Ruler bisection test) and their completion times. Explanatory variables will be age, gender, level of qualification, hand used and laterality.

If no significant association is found between the explanatory variables and the metrics relating to test results and completion times, a mean score with its 95% confidence interval will be estimated.

If there is a significant association between the explanatory variables and the metrics relating to the test results and their completion times, taking into account the characteristics of the healthy volunteers, a mean score for the metrics associated with its 95% confidence interval will be estimated.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteer attending the neurovascular department of Raymond-Poincaré Hospital
2. Aged between 20 and 89 years
3. Affiliated with a health insurance scheme
4. French-speaking
5. Has freely and knowingly expressed their non-opposition

Exclusion Criteria:

1. Known history of central neurological disease: stroke (ischemic or hemorrhagic), transient ischemic attack, encephalitis, multiple sclerosis, or epilepsy.
2. Medical interview suggesting past central nervous system involvement: history of episodes such as sensorimotor deficits, dysarthria, aphasia, blurred or double vision, or positive symptoms such as visual or sensory hallucinations (e.g., paresthesias).
3. Significant visual impairment - as judged by the examiner - in near vision despite correction, or monocular blindness. Specifically, inability to distinguish the targets with gaps in the example (pre-test) of the Apples Cancellation Test.
4. Abnormal neurological examination:

   1. National Institutes of Health Stroke Scale (NIHSS) score > 0
   2. Pyramidal reflex syndrome (hyperactive deep tendon reflexes with extended reflexogenic zones and spread).
5. Use of substances (alcohol or drugs) within 24 hours prior to the assessment.
6. Presence of cognitive or psychiatric disorders, assessed during the inclusion interview and neurological examination, at the examiner's discretion.
7. Language barrier or aphasia, assessed during the inclusion interview and neurological examination, at the examiner's discretion.
8. Participant under legal protection (guardianship, curatorship, or legal safeguard).

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2026-01-07 (Actual); Primary Completion 2027-01-07 (Estimated); Study Completion 2027-01-07 (Estimated)

PRIMARY OUTCOMES:
To establish average scores for healthy French-speaking volunteers without central neurological disorders on the Apples Cancellation Test (from the BCoS), using French-translated administration and scoring instructions | 12 months
  The average scores for healthy French-speaking volunteers without central neurological disorders on the Apples Cancellation Test (from the BCoS), using French-translated administration instructions.
  The number of the box in which the first crossed-out apple is located, the total performance, the spatial asymmetry score (egocentric neglect), the object asymmetry score (allocentric neglect) and the passing time, in seconds.

SECONDARY OUTCOMES:
To establish average scores for healthy French-speaking volunteers without central neurological disorders on the simplified Comb and Razor Test, using French-language administration instructions | inclusion
  The average scores for healthy French-speaking volunteers without central neurological disorders on the simplified Comb and Razor Test, with French-language administration instructions.
To establish average scores for healthy French-speaking volunteers without central neurological disorders on the Peg Test, according to their age, sex, and level of occupational qualification. | inclusion
  The average scores for healthy French-speaking volunteers without central neurological disorders on the Peg Test, according to their age, sex, and level of occupational qualification.
To establish average scores for healthy French-speaking volunteers without central neurological disorders on the 30 cm blind line bisection test using an architect's ruler, according to their age, sex, and level of occupational qualification. | inclusion
  The average scores for healthy French-speaking volunteers without central neurological disorders on the 30 cm blind line bisection test using an architect's ruler, according to their age, sex, and level of occupational qualification.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Raymond Poincarré, Garche, France

IPD SHARING:
Plan to Share IPD: No